CLINICAL TRIAL: NCT03435159
Title: Comparison the Effects of Manual and Instrumental Chiropractic Spinal Manipulation on Vertebrobasilar and Internal Carotis Arteries in Healthy Population
Brief Title: Effects of Spinal Manipulation on Vertebrobasilar and Internal Carotis Arteries in Healthy Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Burcu Özdemir Kocabey, PhD student, Physical Therapist, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: BahcesehirUni
Record Dates: First submitted 2018-01-03; First posted 2018-02-15 (Actual); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Vertebral Artery Dissection, Traumatic; Neck Pain
Keywords: Chiropractic, Manipulation, Vertebrobasilar Artery
MeSH Terms: conditions — Vertebral Artery Dissection; Neck Pain | interventions — Ultrasonography, Doppler

STUDY DESIGN:
Intervention Model Description: 30 participants were divided into 2 groups. In the first group, participants were applied manual chiropractic manipulation, and in the second group, participants were applied instrumental chiropractic manipulation.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Chiropractic Spinal Manipulation (Experimental): Demographic informations, pain, previous trauma, diseases, current medicine, past surgical operations, pregnancy, smoking use and cervical artery dissection history in family are questioned. Cervical flexion, extension, right and left rotations, right and left lateral flexions are measured by physiotherapist, in sitting position and with goniometer.Upper extremity muscle strength was measured with manual muscle testing in sitting position by physical therapist. The muscles innervated by C4, C5, C6, C7, C8 and T1 cervical nerves were examined bilaterally. Cervical foraminal compression test was used to eliminate cervical root compression.Vertebrobasilar artery was assessed by premanipulative vertebrobasilar insufficiency test.Neck Disability Index was used to evaluate the functional neck status of the participants. After all assessments, participants who were eligible for this study were undertaken Doppler Ultrasonography before and after manual manipulative intervention.
  Interventions: Diagnostic Test: Doppler Ultrasonography; Procedure: Manual Chiropractic Spinal Manipulation
- Instrumental Chiropractic Spinal Manipulation (Experimental): The same assessments were applied to determine the eligibility of participants for this study. After all assessments, participants who were eligible for this study were undertaken Doppler Ultrasonography before and after instrumental manipulative intervention.
  Interventions: Diagnostic Test: Doppler Ultrasonography; Device: Instrumental Chiropractic Spinal Manipulation

INTERVENTIONS:
Diagnostic Test: Doppler Ultrasonography — GE LOGIQ S8 ultrasound machine was used to measure blood flow parameters in right and left a. carotis communis, a. carotis interna and a. vertebralis. All vessels were examined in the axial plane through their traces in the B-mode with a C6-15 MHz curvilinear matrix probe. Flow patterns and directions of vessels were then examined with Colour Doppler and it was determined whether there was any stenosis. Intimal thickness of a. carotis communis was measured by spectral doppler method. Measurements were recorded by visualizing the CCA at the supraclavicular level, the ICA carotid sinus (C4 level), and the VA at the V2 segment (C3-4 level), with less angle at 60 degrees. All measurements before and after the application were made at the same level. Immediately after manipulation, blood flow parameters were recorded as numerical data by the same physician again with Doppler USG of the relevant arteries.
Procedure: Manual Chiropractic Spinal Manipulation — Manipulation procedures were applied to C1 or C2 (atlas and axis) vertebrae once in each participant. The application to which vertebrae were applied was determined by the palpation method applied by the physiotherapist. Manual chiropractic manipulation for C1 vertebra was applied in sitting position, using the "digit / atlas pull" technique. This technique is applied with the contact of practitioner's middle finger to the posterior part of transverse process of atlas, and generate a rotation force between C1 and C2 vertebrae.
  The procedure was applied to C2 vertebra using the "index / facet push" technique in the supine position. This technique places pushing force in the direction of rotation between the C2-C3 vertebrae, placing the practitioner's index finger in contact with the posterior surface of the C2 facet joint.
  Arms: Manual Chiropractic Spinal Manipulation
Device: Instrumental Chiropractic Spinal Manipulation — Activator technique was applied to C1 or C2 (atlas and axis) vertebrae once in each participant. The application to which vertebrae were applied was determined by the palpation method applied by the physiotherapist. Instrumental spinal manipulation was applied with Activator V chiropractic instrument. For C1 vertebra, the procedure was applied in supine position, by placing the Activator device horizontally on the participant's atlas transverse process of the affected side and applying a pushing force in the medial direction.
  For C2 vertebra, the procedure was applied in prone position, by placing the Activator device in the relevant C2 pedicle-lamina junction of the participant's affected side and applying a pushing force in the anterior, superior and mild medial direction of movement of the facet joint.
  Other Names: Activator technique
  Arms: Instrumental Chiropractic Spinal Manipulation

SUMMARY:
After lumbar pain, neck pain is the most common cause of patients needing chiropractic care; the second most common cause of spinal manipulation use (1). Manipulation and mobilization are commonly used by chiropractors, osteopaths and manipulative physiotherapists in the treatment of neck pain. Many studies show that the Activator instrument is also used for this purpose in the chiropractic profession (2) There are several published case reports that relate to neck manipulation to vertebral artery dissection and stroke. The prevailing theory is that the neck extension and / or rotation may damage the vertebral artery in the foramen transversarium, especially at the C1-C2 level (2). However, most cases of extracranial vertebral artery dissection are thought to be spontaneous (3).

In the literature, there have been no studies investigating the effects of instrument-assisted spinal manipulation on vertebrobasilar and internal carotis arteries. the aim of this study to compare the effect of manual and instrumental spinal manipulation on blood flow parameters of vertebrobasilar and internal carotis arteries on healthy persons which have mechanical neck pain and asymptomatic in vertebrobasilar insufficiency test.

ELIGIBILITY:
Inclusion Criteria:

* Being between 20-40 years of age
* Having non-specific mechanical neck pain for more than 3 months with symptoms provoked by neck postures, movements, or palpation
* Willingly participating to the study
* Signing the confirmation form.

Exclusion Criteria:

* Spinal root compression (radiculopathy)
* Neurological symptoms like weakness and numbness in extremities and face, uncontrolled movements, abnormal gait, dizziness, undefined nausea/vomiting, swallowing and speaking difficulties
* Acute inflammatory disease
* Spontaneously vertebral artery dissection in family
* Tested positive in premanipulative vertebrobasilar artery insufficiency test
* Being on anticoagulant and antiaggregant medication.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-02-17 (Actual); Primary Completion 2017-04-28 (Actual); Study Completion 2017-04-28 (Actual)

PRIMARY OUTCOMES:
Change in Peak Systolic Velocity (PSV) | 1 minute
  cm/s, measured in each group
Change in End Diastolic Velocity (EDV) | 1 minute
  cm/s, measured in each group
Change in Resistive Index (RI) | 1 minute
  The Formula: RI = (PSV- EDV) / PSV, it has no unit, measured in each group
Change in Volume Flow (VF) | 1 minute
  ml/min, measured only for right and left vertebral arteries

CONTACTS AND LOCATIONS:
Locations (1):
- Maslak Acıbadem Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Gemmell H, Miller P. Relative effectiveness and adverse effects of cervical manipulation, mobilisation and the activator instrument in patients with sub-acute non-specific neck pain: results from a stopped randomised trial. Chiropr Osteopat. 2010 Jul 9;18:20. doi: 10.1186/1746-1340-18-20. PMID 20618936
- [Background] Gemmell H, Miller P. Comparative effectiveness of manipulation, mobilisation and the activator instrument in treatment of non-specific neck pain: a systematic review. Chiropr Osteopat. 2006 Apr 19;14:7. doi: 10.1186/1746-1340-14-7. PMID 16623934
- [Background] Cassidy JD, Boyle E, Cote P, He Y, Hogg-Johnson S, Silver FL, Bondy SJ. Risk of vertebrobasilar stroke and chiropractic care: results of a population-based case-control and case-crossover study. Spine (Phila Pa 1976). 2008 Feb 15;33(4 Suppl):S176-83. doi: 10.1097/BRS.0b013e3181644600. PMID 18204390